### **COVER PAGE**

NJPAG PREIS STUDY PROTOCOL

Protocol ID: NJPAG12131922E

ClinicalTrials.Gov ID: NCT05320666

May 30th, 2023

### Table of Contents

| Introduction | 4 |
|----------------------------------------------------------|----|
| Intervention Activities | 4 |
| Logic Model | 5 |
| Target Population | 6 |
| Impact Evaluation | 6 |
| Impact Evaluation Overview | 6 |
| Research Questions | 6 |
| Study Registration | 8 |
| Conflicts of Interest | 8 |
| Treatment and Comparison Conditions | 8 |
| Treatment Condition | 8 |
| Control/Comparison Condition | 8 |
| Sample Identification, Selection, and Retention | 8 |
| Anticipated Sample Size | |
| Identification and selection of clusters (if applicable) | 9 |
| Identification and selection of individuals | |
| Tracking and Retention of Individuals | |
| Data Collection | |
| Data Collection Plan | |
| Specific Measures, Tools, and Instruments | 14 |
| Anticipated Challenges | |
| Data Sharing/ Data Use Agreements | |
| Analysis | |
| Analysis Plan | |
| Contrasts | |
| Subgroups (optional) | |
| Minimum Detectable Effect for Planned Sample | |
| Timeline | |
| Approvals and Data Security | |
| Plan for IRB Approval | |
| Plan for federal Wide Assurance | |
| Data Security & Privacy | |
| Evaluation Roles and Responsibilities | 20 |
| Appendix A. Logic Model | 21 |
| Appendix B. Contrast Table | |
| Appendix C: Parental Written Notice | |
| Appendix D: Enrollment Form | |
| Appendix E: Survey | |
| YOUTH ASSENT FORM | |
| DEMOGRAPHICS | 39 |
| PROGRAM SATISFACTION QUESTIONS | 40 |
| COMMUNICATION SKILLS | 40 |
| DATING CHOICES | |
| AWARENESS OF RELATIONSHIP SAFETY | |
| KNOWLEDGE OF SEXUAL RISKS | |
| SKILLS TO RESIST PRESSURE (COERCION) TO HAVE SEX | |
| SEXUAL INTIMACY SPECTRUM | |
| SEXUAL INITIATION | |
| INTENTIONS TO ENGAGE IN SEXUAL INTERCOURSE | |

| | 3 |
|------------------------------------|----|
| INTENT TO CONSISTENTLY USE CONDOMS | 47 |
| CONDOM & CONTRACEPTIVE USAGE | 48 |
| GOAL ATTAINMENT | 49 |
| FINANCIAL LITERACY | 49 |
| END OF SURVEY | 50 |

### Introduction

The New Jersey Physicians Advisory Group (NJPAG) previously created the *Yes You Can...Make Smart Choices!* (YYC...MSC!) program with the goal of preventing teen pregnancy and enhancing character development in youth. YYC...MSC! is a fully developed intervention that NJPAG has experience implementing that is grounded in a theoretical framework with promising evidence of effectiveness. However, this intervention has not yet undergone a rigorous evaluation with a control or comparison group. This evaluation aims to conduct a randomized control trial (RCT) to determine the program's effectiveness. This evaluation will focus on the entire PREIS planned intervention, YYC...MSC!. The intervention will be implemented in 10 Newark Public Schools in New Jersey, including Weequahic High School and Newark School of Global Studies. Findings from this study will expand the evidence base on adolescent pregnancy prevention through this innovative program. After the study, findings will be disseminated to encourage program interest, support, and adoption in real-world service systems or communities, including schools.

### **Intervention Activities**

The YYC...MSC! is an 11-lesson curriculum that will be delivered to 9<sup>th</sup> graders in Newark, New Jersey public schools during 40-minute health classes (see Table 1 for content covered in each lesson). The curriculum will be delivered in-person over approximately 2 weeks by NJPAG educators. The goal of the program is to prevent teen pregnancy and enhance character development in youth. The PREIS funding is supporting the implementation and evaluation of the program. Each time an NJPAG educator is in the classroom, they will deliver a single lesson of the curriculum. All NJPAG educators have received internal training for the program; their training includes: (1) studying the curriculum and completing activity/learning pages, (2) practicing teaching to other educator in a mock classroom setting, followed by feedback from the team, (3) observing a seasoned educator teaching the curriculum in its entirety, (4) coteach the curriculum with a seasoned educator, and (5) teaching on their own, with observation. YYC...MSC! is delivered like a traditional classroom curriculum, including lectures and activities, meaning all students in a given classroom will receive the lectures concurrently. The intervention addresses the following adult preparation subjects: parent-child communication, healthy relationships, healthy life skills, adolescent development, and financial literacy.

Table 1. YYC...MSC! Curriculum Lesson Goals

| Lesson | Goal |
|---|---|
| Lesson 1: Truth, Dare, or Consequences? | Students will understand the influences and consequences of sexual activity. |
| Lesson 2: Dare To Be<br>You | Students will understand how others influence their character development and decision-making. |
| Lesson 3: Intimacy | Students will understand intimacy and when to be intimate in relationships. |
| Lesson 4: Relationship<br>Health Part 1 | Students will begin to understand what love is and how to have healthy relationships. |
| Lesson 5: Relationship<br>Health Part 2 | Students will continue to understand what love is and know the difference between a healthy and unhealthy relationship. |

| Lesson 6: Pregnancy | Students will understand pregnancy, how to prevent it, and the consequences of teen pregnancy. |
|---|---|
| Lesson 7: Finances and Future Planning | Students will understand the basics of financial literacy and creating financial goals. |
| Lesson 8: Avoiding<br>Risk | Students will understand HIV/AIDs, STDs/STIs, unintended pregnancy, and how to prevent them. |
| Lesson 9: What Are We Waiting For? | Students will understand the benefits of refraining from sexual activity. |
| Lesson 10: Establishing<br>Healthy Boundaries | Students will understand personal boundaries and how to resist and refuse sexual activity. |
| Lesson 11: Effective<br>Communication | Students will understand and obtain skills for effective communication, including with parents/guardians. |

### Logic Model

See Appendix A for the intervention logic model. Since its inception in 2004, NJPAG has been a non-profit in New Jersey with the goal of addressing the societal problems of teen pregnancy, teen STDs/STIs, and single-parent teen families. To meet this goal, NJPAG has created various curricula to educate youth in New Jersey and beyond, including the YYC...MSC! curriculum for this intervention. NJPAG has a positive, existing relationship with the Newark Public Schools (NPS) Board of Education. As a result of this relationship, NJPAG has the approval to provide the intervention as part of all NPS's 9<sup>th</sup>-grade health classes. Schools with potentially high rates of language barriers were eliminated because the program is only taught in English. After eliminating schools with potentially high rates of language barriers, 10 NPS schools were selected to participate in the evaluation, five control schools, and five treatment schools.

Internally, NJPAG has a Board of Directors, Executive Director, Program Director, and educators. After receiving training, NJPAG educators will go into Newark public high schools to build rapport with the school's teachers, staff, and students and explain the intervention and related processes. Once rapport is built, NJPAG will go to classes and disseminate the written notice form for youth to bring home to parents to inform parents of the program their child/student will receive and give the parents the option to opt their child/student out of the evaluation. Two weeks after the written notice is disseminated, an Educator will go back to the classroom and collect any forms returned by parents who opted their child out of the evaluation. Upon receiving opt-outs, an educator will facilitate the pre-survey. The following school day after the presurvey, the educator will go back to the classroom to begin program delivery, starting with lesson 1 and subsequently teaching a lesson every time they go to the classroom. Each lesson addresses a different topic related to pregnancy prevention and has lesson goals (see Table 1).

We expect all lessons to work together to achieve the program goal. For intermediate outcomes, we expect that treatment school youth, e.g., those that receive the intervention, will report an increase in pregnancy prevention knowledge, skills, and confidence and a decrease in activity that could lead to unwanted pregnancy. We believe this intervention will impact youth who received the program long-term by improving life skills, such as emotional coping and sexual, cognitive, and social health, decreasing incidences of unwanted pregnancy, decreasing incidences of STIs, and enhancing character development.

### **Target Population**

NJPAG has been serving New Jersey public schools for almost two decades. Recently, NJPAG was approved to provide sex education programming to 9<sup>th</sup>-grade health class students in NPS by the Newark Board of Education

The target population is youth in 9<sup>th</sup> grade in urban school districts in the Northeast region without any severe cognitive, mental, or behavioral impairments.

The total population of youth who would receive the intervention is approximately 2,000 students. The average expected age of participants is 14. Consistent with the NPS district student population race/ethnicity breakdown, the expected race/ethnicity breakdown of participants is as follows: Black (38.8%), Hispanic (51.0%), White (8.4%), Asian (< 1%), Native Hawaiian/ Pacific Islander (< 1%), American Indian (< 1%), Unspecified (< 1%).

### **Impact Evaluation**

This study will utilize an RCT design, in which randomization is done at the school level. Ten NPS schools are participating in the evaluation, indicating five treatment and five control schools.

### Impact Evaluation Overview

### **Research Questions**

The intervention being tested is the YYC...MSC! program and the target population are youth in 9<sup>th</sup> grade in urban school districts in the Northeast region without any severe cognitive, mental, or behavioral impairments. The counterfactual condition is business as usual for control schools. The intervention occurs over 11 consecutive school days in health classes.

The *primary research question* is, "What is the effect of the 2-week YYC...MSC! program on 9th grade students in Northeast urban school districts' reports of engaging in sexual intercourse 12-months after the presurvey compared to those that do not receive the program?" The outcome for the primary research questions is sexual intercourse in the last 3 months and the domain is sexual activity.

There are 12 secondary research questions; including (1) What is the effect of the 2-week YYC...MSC! program on 9th grade students in Northeast urban school districts' reports of engaging in oral sex compared to those that do not receive the program? [domain: sexual activity, outcome: oral sex], (2) What is the effect of the 2-week YYC...MSC! program on 9th grade students in Northeast urban school districts' reports of intent to engage in sexual activity, outcome: intent to engage in sexual activity], (3) What is the effect of the 2-week YYC...MSC! program on 9th grade students in Northeast urban school districts' reports intent to consistently use contraception compared to those that do not receive the program? [domain: sexual risk avoidance intent, outcome: consistent contraception use], (4) What is the effect of the 2-week YYC...MSC! program on 9th grade students in Northeast urban school districts' reports of having unprotected sex compared to those that do not receive the program? [domain: sexual risk avoidance, outcome: unprotected sex], (5) What is the effect of the 2-week YYC...MSC! program on 9th grade students in Northeast urban school districts' reports of

increased financial literacy compared to those that do not receive the program?" [domain: life skills, outcome: financial literacy], (6) What is the effect of the 2-week YYC...MSC! program on 9th grade students in Northeast urban school districts' knowledge of HIV/STDs/STIs compared to those that do not receive the program? [domain: sexual health knowledge, outcome: knowledge of HIV/STIs/STDs], (7) What is the effect of the 2-week YYC...MSC! program on 9th grade students in Northeast urban school districts' reports of their ability to resist negative pressures to have sex compared to those that do not receive the program? [domain: sexual risk avoidance skills, outcome: skills to resist pressure], (8) What is the effect of the 2-week YYC...MSC! program on 9th grade students in Northeast urban school districts' reports of future orientation and setting life goals compared to those that do not receive the program? [domain: life skills, outcome: goal setting], (9) What is the effect of the 2-week YYC...MSC! program on 9th grade students in Northeast urban school districts' reports of healthy life skills compared to those that do not receive the program? [domain: life skills, outcome: healthy life skills], (10) What is the effect of the 2-week YYC...MSC! program on 9th grade students in Northeast urban school districts' knowledge of healthy relationships compared to those that do not receive the program? [domain: life skills, outcome: healthy relationships], (11) What is the effect of the 2-week YYC...MSC! program on 9th grade students in Northeast urban school districts' increased communication skills compared to those that do not receive the program? [domain: life skills, outcome: communication], and (12) What is the effect of the 2-week YYC...MSC! program on 9th grade students in Northeast urban school districts' engaging in sexual intercourse 3-months after the pre-survey? [domain: sexual activity, outcome: sexual intercourse in the last 3-months].

| Research Question / Hypothesis | Primary<br>or<br>Secondary? | Domain | Outcome |
|---|---|---|---|
| What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' reports ofthat do not receive the program? | | | |
| RQ 0 engaging in sexual intercourse 12-months after the presurvey? | Primary | Sexual Activity | Sexual Intercourse in the last 3-months |
| RQ 1 engaging in oral sex? | Secondary | Sexual Activity | Oral sex |
| RQ 2intent to engage in sexual activity? | Secondary | Intent to Engage in Sexual Activity | Intent to Engage in Sexual Activity |
| RQ 3 their intent to consistently use contraception? | Secondary | Sexual Risk Avoidance<br>Intent | Consistent<br>Contraception Use |
| RQ 4 having unprotected sex? | Secondary | Sexual Risk Avoidance | Unprotected Sex |
| RQ 5 increased financial literacy? | Secondary | Life Skills | Financial Literacy |
| RQ 6 knowledge of HIV/STDs/STIs? | Secondary | Sexual Health Knowledge | Knowledge of HIV/STI/STDs |
| RQ 7 their ability to resist negative pressure to have sex? | Secondary | Sexual Risk Avoidance<br>Skills | Skills to Resist<br>Pressure |
| RQ 8 future orientation and setting life goals? | Secondary | Life Skills | Goal Setting |
| RQ 9 healthy life skills? | Secondary | Life Skills | Healthy Life Skills |

| RQ 10 knowledge of healthy relationships? | Secondary | Life Skills | Healthy Relationships |
|---|---|---|---|
| RQ 11 communication skills? | Secondary | Life Skills | Communication |
| RQ 12 engaging in sexual intercourse 3-months after the presurvey? | Secondary | Sexual Activity | Sexual Intercourse in the last 3-months |

### Study Registration

The evaluation will be registered at clinicaltrials.gov.

### Conflicts of Interest

There are no conflicts of interest.

Treatment and Comparison Conditions

### **Treatment Condition**

The intervention/treatment participants in the treatment condition will be exposed to NJPAG's YYC...MSC! program. The program is designed to be delivered five days a week for two weeks and contains 11 lessons (see Table 1 for lessons and goals).

### Control/Comparison Condition

The control schools were randomly selected out of a list of eligible schools (a total of 10) in the Newark Public School system. Control schools will receive their health class as "business-as-usual" with no additional programming. There is no other place that provides the YYC...MSC! program in which participants could receive programming or information. Also, there are no future plans to provide the control group with the intervention. To our knowledge, there is no other similar programming operating in the Newark Public School area.

### Sample Identification, Selection, and Retention

The YYC... MSC! program is approved as the Newark Board of Education sexual education curriculum. All 9<sup>th</sup> graders in the ten selected NPS schools will be asked to participate in the evaluation. Newark public schools with a high percentage of English Language Learners (ELL) students since the program is only provided in English. Participants will be identified by being in a school that is randomly assigned to be a treatment school. Ninth graders in participating NPS treatment schools will receive the YYC...MSC! program.

Program attrition is predicted to be minimal, given it is a school-based program. However, attrition is likely for students who move out of the district or to another school within the district. To try to reach students that move, we are collecting contact information (phone number and personal email address) on our enrollment form. Cluster-level attrition is predicted to be unlikely given the rapport NJPAG has previously built with the Newark Public Schools individually and as a district.

### **Anticipated Sample Size**

We currently have ten public schools that are engaged in this study, five that will be randomly assigned to the treatment group and five that will be randomly assigned to the control group. On average, there are four health classes in each school, each of which has approximately 25 students. Therefore, each year we will enroll approximately 1,000 students in the study ( $25 \times 4 \times 10 = 1,000$ ); 500 in the treatment group and 500 in the control group. Unless we are able to recruit more schools (we are currently having conversations with several charter schools in the Newark School District), we anticipate having to run the study for two full years, in order to meet the sample size requirements needed to achieve adequate power. We will then have 2,000 students enrolled in the study (1,000 in the treatment group and 1,000 in the control group).

### Identification and selection of clusters (if applicable)

The 10 eligible Newark Public Schools were selected as clusters. There is only one exclusionary criterion for schools, and that is a high percentage of ELL students because the program is only offered in English. Given the buy-in from the Newark Board of Education, recruiting schools is not anticipated to be a problem. NJPAG has started building rapport with the department chairs at each of the participating schools and providing a \$1,000 incentive for their cooperation. The level of randomization is at the school-level, meaning we will randomly assign each of the 10 schools to either treatment or control. Random assignment will be conducted using a random number generator from 0-1 in Excel. After generating random numbers, the ten schools will be ordered based on their number assignment and the five with the smallest number will be assigned control and the five with the highest number will be assigned treatment. All students included in the impact analysis will be students of the participating schools prior to random assignment. Students will be notified of their schools' random assignment after the parental written notice is distributed and enrollment is completed.

### Identification and selection of individuals

Youth served and recruited will be limited to 9<sup>th</sup> graders from health classrooms at the NPS sites participating in this program who do not have severe cognitive, mental, or behavioral impairments. Students with an Individual Education Plan (IEP) who are in a restricted placement due to such issues will not be able to participate in the program as they will not be a part of the mainstream classrooms where the program will take place. Students with an IEP who are placed in regular classroom settings (i.e., mainstreamed) will be included in the program.

New Jersey law only requires passive parental consent to be obtained, using a written notice about the evaluation provided to students to bring home with an option for parents to sign the notice to opt their child/student out of the evaluation. If parents wish to opt their child/student out of the evaluation, the child will still receive the program because it is the Newark Board of Education-approved sexual education curriculum treatment group health classes. When the Educator goes back to the classroom to pre-survey, they will collect any 'opt-out' notices and survey only those students whose parents have not elected to 'opt-out' their child.

Ineligible students include students with IEP who are in a restricted placement and students that bring back 'optout' written notices. Since we are using the same form for treatment and control schools (making it unclear to parents what group their child is in), we do not expect differences in opt-out rates between treatment and control schools.

Given NJPAG's relationship with the Newark Board of Education, recruitment of schools is not expected to be challenging. NJPAG will contact each of the eligible schools to communicate about the program, program delivery, and the timeline. Schools will be randomized and maintain their randomization category for the entirety of the evaluation for pragmatic reasons (e.g., NJPAG-school communication, building rapport, etc.). After randomization, NJPAG Educators will go into schools to tell the students about the evaluation. Students at this time will not know if they are receiving the program. Following that, students are told to bring home the

written notice and provide it to their parents for the option to opt out of the evaluation. Additionally, health class teachers are given an incentive (\$25 gift card) per participating health class to show the program's appreciation for their cooperation For each-school, the timeline goes as follows: Educator goes into school and health classes to disseminate the written notice for youth to bring home to their parents, the Educator comes back 2 weeks later to pre-survey all participating youth, the next school day the Educator comes back to start the program and consistently teaches a lesson for the next 11 school days, the next school day a different Educator goes into the school health classes to collect post-survey data, 3-months after the pre-survey date a different Educator goes into the school health classes to collect follow-up data, and 12-months after the pre-survey date a different Educator goes into the school health classes to collect follow-up data.

For the current study, no program enrollment is necessary because the NPS Board of Education approved the YYC...MSC! program as a designated sexual health curriculum for 9<sup>th</sup> graders. Therefore, all students in NPS treatment sites will be automatically enrolled in the program; but parents can opt their child out of the evaluation. Evaluation enrollment will be obtained via parental opt-out forms.

The process for each cohort is the following: NJPAG Educator goes into school, tells youth about the program and evaluation, and disseminates parental written notices.

- (1) Educators collect any 'opt-out' notices that were returned.
- (2) All participating students take the pre-survey.
- (3) Students receive full YYC...MSC! Programming.
- (4) All participating students take the post-survey.

Follow-Up

- (5) Participating students take a follow-up survey 3-months after the pre-survey date.
- (6) Participating students take a follow-up survey 12 months after the pre-survey date.

### Tracking and Retention of Individuals

Because the YYC...MSC! program was approved by the Newark Board of Education as a sex education program for NPS 9<sup>th</sup> graders required health classes; program dosage and attendance will be consistent with students' health class attendance. For follow-up data collection, NJPAG Educators will go back into the school building and pull participating students from their classes to participate in follow-up surveys. If a given participant is not there when the NJPAG Educator goes back to the school to collect follow-up data, we will communicate with the school district contact to attempt to locate the participating students to survey them at their new school. If a participating student moves out of the Newark school district, we will contact them via phone or email and ask them to participate in the survey. The anticipated response rate for each round of data collection is as follows: pre-survey (95%), post-survey (85%), three months (80%), and 12 months (70%). Participating students will receive \$0 for completing the pre-survey, \$20 after completing the post-survey, \$30 after completing the 3-month follow-up survey, and \$40 after completing the 12-month follow-up survey.

### **Data Collection**

### Data Collection Plan

Participants in the treatment group will be determined to have completed their engagement in the intervention if they received 80% of the program lessons (e.g., 9 out of 11). The data collection window for each time point is two weeks. The data collection window will be managed by reviewing participants' timestamp (e.g., the time and date they started the survey) on their survey completion. There are no costs associated with measures because they were all created for this project specifically.

The timing of data collection for the pre-survey is before the first lesson is administered, approximately 2 weeks after disbursing the written notice for students to bring home to their parents. The post-survey is collected immediately following the completion of the program. The 3-month follow-up survey is collected 3-months from the pre-survey date. The 12-month follow-up is collected 12-months from pre-survey.

Corresponding survey questions for all research questions will be collected at all timepoints. In the below table, data collection times in which the data will be collected but not analyzed is characterized by a black X. Orange Xs in the below table represent the timepoint in which we will analyze the data for the research question.

*Note*: The following are constants in the below table for each research question:

Data source (and measures): Self-report surveys by student participants

Sample: All treatment and control group participants Party responsible for data collection: NJPAG educators Data collection method: Electronic surveys via Alchemer

| | Data Collection Timing | | | |
|---|---|---|---|---|
| Impact research question | Pre-<br>Survey/<br>Baseline | Post-Survey | 3-Month<br>After Pre-<br>Survey | 12-Month<br>After Pre-<br>Survey |
| RQ 0 – Primary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' reports of engaging in sexual intercourse 12-months after the pre- survey compared to those that do not receive the program? | X | X | X | X |
| RQ 1 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' reports of engaging in oral sex compared to those that do not receive the program? | X | X | X | X |
| RQ 2 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' reports of intent to engage in sexual activity compared to those that do not receive the program? | X | X | X | X |
| RQ 3 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' reports intent to consistently use contraception compared to those that do not receive the program? | X | X | X | X |

| | Data Collection Timing | | | |
|---|---|---|---|---|
| Impact research question | Pre-<br>Survey/<br>Baseline | Post-Survey | 3-Month<br>After Pre-<br>Survey | 12-Month<br>After Pre-<br>Survey |
| RQ 4 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' reports of having unprotected sex compared to those that do not receive the program? | X | X | X | X |
| RQ 5 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' increased financial literacy compared to those that do not receive the program? | X | X | X | X |
| RQ 6 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' knowledge of HIV/STDs/STIs compared to those that do not receive the program? | X | X | X | X |
| RQ 7 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' reports of their ability to resist negative pressures to have sex compared to those that do not receive the program? | X | X | X | X |
| RQ 8 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' reports of future orientation and setting life goals compared to those that do not receive the program? | X | X | X | X |
| RQ 9 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' reports of healthy life skills compared to those that do not receive the program? | X | X | X | X |
| RQ 10 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' knowledge of healthy relationships compared to those that do not receive the program? | X | X | X | X |

| | Data Collection Timing | | | |
|---|---|---|---|---|
| Impact research question | Pre-<br>Survey/<br>Baseline | Post-Survey | 3-Month<br>After Pre-<br>Survey | 12-Month<br>After Pre-<br>Survey |
| RQ 11 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' increased communication skills compared to those that do not receive the program? | X | X | X | X |
| RQ 12 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' engaging in sexual intercourse 3-months after the pre-survey? | X | X | X | X |

| Domain | Outcome | Measure | Rationale for Selection |
|---|---|---|---|
| Sexual<br>Activity | Sexual<br>Intercourse in<br>the last 3-<br>months | 1-item measure asking participants how many times they engaged in sexual intercourse in the past 3-months recoded to a dummy variable (1 = had sex in the last 3-months, 0 = did not have sex in the last 3-months) | Reducing sexual intercourse rates in youth, to, in turn, reduce teen pregnancy, is the primary goal of this intervention. |
| Sexual<br>Activity | Oral sex | 8-item Sexual Intimacy Spectrum scale with a 5-point frequency scale Two 1-item measures asking participants if they ever engaged in oral sex if so, how many times have they done it in the past 3-months | Following the success sequence, the program teaches youth that engaging in sexual activity before they are ready and have hit life milestones can have unwanted consequences. |
| Intent to<br>Engage in<br>Sexual<br>Activity | Intent to Engage in Sexual Activity | 8-item Sexual Initiation scale with a 5-point success sequence response scale 5-item Intentions to Engage in Sexual Intercourse scale with a 6-point Agree scale | Following the success sequence, the program teaches youth that engaging in sexual activity before they are ready and have hit life milestones can have unwanted consequences. |
| Sexual Risk<br>Avoidance<br>Intent | Consistent<br>Contraceptive<br>Use | Two 1-item measures asking: "If you have sexual intercourse tomorrow, will you make sure a condom is used?" & "If you have sexual intercourse tomorrow, will you make sure birth control is used?" Both questions use the same 5-point response scale: "Yes; No; Only if my partner agrees; I don't know/I'm not sure; This question does not apply to me because I do not plan to have sexual intercourse soon" | Contraceptive use is important because the intervention teaches youth about pregnancy prevention. It is important to assess all students' intention to use contraception if they have sexual intercourse because the program is a pregnancy prevention program. |
| Sexual Risk<br>Avoidance | Unprotected<br>Sex | Four 1-item measures asking if youth or their partner have used the following methods in the last month and what they intend to use in the future: condoms, pull-out method, birth control, other contraceptives If youth indicate that they have engaged in sexual intercourse at some time in the last 3-months, they will respond to two 1-item | It is important to assess all student's rates of unprotected sex because the program is a pregnancy prevention program. |

| | T | T | 13 |
|---|---|---|---|
| | | measures & one 2-item measure asking if they have used conceptive during sexual intercourse | |
| | | In the <b>past 3 months</b> (90 days), how many times did you or your partner use a condom when engaging in sexual intercourse? Response: 0-10+ | |
| | | In the <b>past 3 months</b> (90 days), how many times did you or your partner use the pull-out method when engaging in sexual intercourse? Response: 0-10+ Or I don't know what this is. | |
| | | In the past 3 months, have you or your partner used either of the following methods to prevent pregnancy: 1. Birth control pills 2. Other forms of contraceptive methods, not including a condom (e.g., shot, patch, IUD, etc.). Response options: Yes, No, Unsure | |
| Life Skills | Financial<br>Literacy | 6-item Financial Literacy scale – 3 items are true/false, and the other 3 are strongly disagree-strongly agree | Financial literacy is a lesson in the YYCMSC! program. |
| Sexual<br>Health<br>Knowledge | Knowledge of<br>HIV/<br>STDs/STIs | 7-item Knowledge of Sexual Risks scale with True/False/Unsure response scale | The intervention teaches a lesson on HIV/STD/ STIs and how to prevent them. |
| Sexual Risk<br>Avoidance<br>Skills | Skills to Resist<br>Pressure | 6-item Skills to Resist Pressure (Coercion) to Have Sex scale with a 5-point Confidence response scale | There are multiple lessons in<br>the intervention that teach<br>participants about negotiating<br>sexual risk avoidance and not<br>falling for pressures to have<br>sex. |
| Life Skills | Goal Setting | 5-item Goal Attainment scale with a 6-point Agree response scale | In addition to pregnancy prevention, the program encourages and teaches youth to think about their life goals and how, if they were to get pregnant, that could negatively impact their goals. |
| Life Skills | Healthy Life<br>Skills | Combination of all scales except Financial Literacy | An overall theme of the intervention is increasing healthy life skills (e.g., |

| | | | emotional, cognitive, and social) for youth. |
|---|---|---|---|
| Life Skills | Healthy<br>Relationships | 6-item Awareness of Relationship Safety scale with a 6-point strongly disagreestrongly agree response scale 7-item Dating Choices scale with a 4-point Likelihood response scale | The intervention teaches youth about healthy relationships for their age and when to know if they are in an unhealthy relationship. |
| Life Skills | Communication | 7-item Communication Scale with a 5-point Confidence scale | The intervention teaches youth communication skills. |

*Note*: The following are constant for all outcomes:

Intended participants: Student participants

Psychometric Information: All scales will go through reliability testing using pilot study data. Citations: N/A – All measures were adapted or created specifically for this project. Scales that were adapted for this project were adapted from AMTC created and unpublished scales for other AMTC clients. Validity and reliability will be conducted after data collection.

### **Anticipated Challenges**

All data is self-report through surveys; however, sexual behavioral questions may make youth uncomfortable, so we predict that this data may be most challenging to collect. To mitigate this, we have ordered the survey to go from the least uncomfortable topics to the most uncomfortable topics in hopes of "building up" to the most uncomfortable topics. Another anticipated challenge is following up with students for the follow-up surveys, the current strategies for this include (1) going back to the schools to survey youth, so if they are in attendance at school, they will take the survey, and if the students no longer attend that school or are not present on follow-up survey dates (2) we have collected their phone number and email to send them a link to the survey to complete the survey. Most participating youth will be surveyed as a group when Educators go back to classrooms; however, youth that has left the district will be contacted via email and/or phone to find a way to provide them with a survey link that they can complete within the two- week survey completion window. Youth that receive the survey via email will receive reminder emails to complete the survey.

### Data Sharing/ Data Use Agreements

N/A – there are no data/sharing agreements for the project.

### Analysis

### Analysis Plan

All analyses will be conducted using SPSS. Outliers will be identified as three standard deviations above the mean and removed from the data. When appropriate, missing data will be handled by using mean imputation. This will only occur when feasible. For example, if participants have skipped over a subset of items on a particular measurement scale, we can use mean imputation for their missing data. However, we will be unable to use mean imputation for behavioral outcomes that are only measured by a single item. Participant data will

be utilized for analyses if they completed 75% of scale items within a given scale. We will use categorial data analysis, such as logistic regression, to analyze any outcomes that are measured using a single item. We will use multiple regression to analyze outcomes that are measured using multiple items. Baseline/pre-survey data will be used as a covariate in all models. Level 1 covariates include race, gender, age, and sexual orientation. There is one Level 2 covariate, school size.

Contrasts

See Appendix B.

Subgroups (optional)

We will analyze data by demographic groups, including gender identity, sexual orientation, and race to explore different programmatic impacts and experiences based on these categories.

### Minimum Detectable Effect for Planned Sample

### **Power Analysis**

Our evaluation is a two-level simple cluster random assignment design. Level 1 (unit of analysis) is individual students, and Level 2 (unit of assignment) is schools. The alpha level is set to 0.05 following conventional statistics, as we only have one primary research question. The test will be a two-tailed test to assess for any positive or negative change resulting from the program. Following conventional statistics, Power is set to 0.80. Rho (ICC) is set to 0.02 because we expect little variable in outcome between clusters. We will randomly assign the ten schools to treatment and control, resulting in five schools in treatment and five in control (P = 0.50). Following suggestions from the Program Officer, we set our  $R^2$  values to 0.20. We will have one Level 2 covariate, e.g., school size. We expect 150 participating students in each school. We currently have ten guaranteed schools in the study but are exploring adding more.

| Model 3.1: MDES Calculator for Two-Level Cluster Random Assignment Design (CRA2_2)— Treatment at Level 2 | | |
|---|---|---|
| Assumptions Comments | | |
| Alpha Level (α) | 0.05 | Probability of a Type I error |
| Two-tailed or One-tailed Test? | 2 | |
| Power (1-β) | 0.80 | Statistical power (1-probability of a Type II error) |
| Rho (ICC) | 0.02 | Proportion of variance in outcome that is between clusters |
| P | 0.50 | Proportion of Level 2 units randomized to treatment: $J_T / (J_T + J_C)$ |
| ${\bf R_1}^2$ | 0.20 | Proportion of variance in Level 1 outcomes explained by Level 1 covariates |
| $\mathbb{R}_2^{\ 2}$ | 0.20 | Proportion of variance in Level 2 outcome explained by Level 2 covariates |
| g* | 2 | Number of Level 2 covariates |
| n (Average Cluster Size) | 150 | Mean number of Level 1 units per Level 2 cluster (harmonic mean recommended) |
| J (Sample Size [# of Clusters]) | 10 | Number of Level 2 units |
| M (Multiplier) | 3.35 | Computed from T <sub>1</sub> and T <sub>2</sub> |
| T <sub>1</sub> (Precision) | 2.45 | Determined from alpha level, given two-tailed or one-tailed test |
| T <sub>2</sub> (Power) | 0.91 | Determined from given power level |
| MDES | 0.309 | Minimum Detectable Effect Size |

### Timeline

| Impact Evaluation Activity | Start Date | End Date |
|---|---|---|
| IRB submission | 3/1/2023 | 4/1/2023 |
| Registering the study | 4/1/2023 | 5/1/2023 |
| COHORT 1 – FALL 2023 | | |
| Baseline/pre-survey data collection | 9/25/2023 | 10/2/2023 |
| Post-survey data collection | 10/2/2023 | 10/16/2023 |
| 3-month follow-up data collection | 1/2/2024 | 1/16/2023 |
| 12-month follow-up data collection | 9/25/2024 | 10/2/2024 |
| COHORT 2 – SPRING 2024 | | |
| Baseline data collection | 3/1/2024 | 3/15/2024 |
| Post-survey data collection | 3/15/2024 | 3/30/2024 |
| 3-month follow-up data collection | 6/1/2024 | 6/15/2024 |
| 12-month follow-up data collection | 3/1/2025 | 3/15/2025 |
| COHORT 3 – FALL 2024 | COHORT 3 – FALL 2024 | |
| Baseline data collection | 9/25/2024 | 10/2/2024 |
| Post-survey data collection | 10/2/2024 | 10/16/2024 |
| 3-month follow-up data collection | 1/1/2025 | 1/15/2025 |

| Impact Evaluation Activity | Start Date | End Date |
|------------------------------------|------------|------------|
| 12-month follow-up data collection | 9/25/2025 | 10/2/2025 |
| COHORT 4 – SPRING 2025 | | |
| Baseline data collection | 3/1/2025 | 3/15/2025 |
| Post-survey data collection | 3/15/2025 | 3/30/2025 |
| 3-month follow-up data collection | 6/1/2025 | 6/15/2025 |
| 12-month follow-up data collection | 3/1/2026 | 3/15/2026 |
| ANALYSIS & DISSEMINATION | | |
| Analysis | 3/15/2026 | 5/15/2026 |
| Reporting | 5/15/2026 | 8/15/2026 |
| Dissemination | 8/15/2026 | 12/31/2026 |

### Approvals and Data Security

### Plan for IRB Approval

We have obtained the Biomedical Research Alliance of New York Institutional Review Board (BRANY IRB) approval. All staff, including evaluators and NJPAG Educators, have received human subjects protection training.

### Plan for federal Wide Assurance

The FWA for the current study was obtained from Research Analytics Consulting and is FWA00031511 (Expiration date: July 21<sup>st</sup>, 2026).

### Data Security & Privacy

Survey data collection will be captured electronically via Alchemer.com, ensuring the quality and security of both data collection and data storage. Individual-level federal reporting and tracking data is captured and stored on AMTC & Associates Online Participant Tracking System (OPTS) (further security information can be found below). Data collectors are trained in the protection of human subjects and best practices for successful data collection.

Electronic surveys will be collected using online surveys from Alchemer.com. Alchemer is committed to ensuring the quality and security of its data collection software and has robust monitoring software used to monitor performance and notify any issues.

All staff working with Personally Identifiable Information (PII) and sensitive data complete training on the program policy and sign a confidentiality form agreeing not to share participant-level PII or sensitive data. Access to data will only be granted to project staff who need access and sign a confidentiality agreement such

as staff responsible for data collection, entry and/or electronic or hard copy transmission; these staff must be trained on and sign the receipt of this policy and confidentiality agreement. Those who may only need limited access will be trained and will sign the receipt of the policy. Limited access to data may include only having access to the necessary data to understand the number of responses for each school, class, and teacher. For example, facilitators may collect attendance data but may not need access to survey data, and yet attendance data may be related to sensitive data. Additionally, identifiable data from surveys will only be available to the analysts tasked with de-identifying the data. Documents containing PII (e.g., completed parent consent forms) will be saved on a secure computer server away from survey data. Data will be de-identified. To link entry, exit, and follow-up surveys, a pseudo-ID will be created by asking the youth for their first and last initials, birth month, and birth date on each survey administered. These individual survey items will be concatenated to create a unique ID for each respondent.

If a data breach occurs, Evaluators will notify NJPAG, pause data collection, identify any vulnerable parties, fix any issues resulting from a breach, and ensure any improperly shared information is deleted.

**Evaluation Roles and Responsibilities** 

| Name | Contact Information | Experience | Organization | Role in<br>Evaluation |
|---|---|---|---|---|
| Peggy<br>Cowan | pcowan@njphysic<br>ians.org | 19 years of experience as the President of NJPAG, previously contributing to program evaluation and managing grants. | NJPAG | President of PREIS Recipient |
| Debbie<br>Marchione | debbie@njphysici<br>ans.org | 10+ years of experience working for NJPAG in a variety of capacities, contributing to program evaluation and managing grants. | NJPAG | Program Director of PREIS program |
| Dr. Cindy<br>M. Walker | cindy@researchan<br>alyticsconsulting.c<br>om | 25+ years of experience conducting research and evaluations with various partners (e.g., community-based organizations, government entities. State and local school districts), including projects related to pregnancy prevention and sexual risk avoidance in youth | Research<br>Analytics<br>Consulting | Leading<br>Evaluator |
| Helena<br>Lucia<br>Swanson | helena@researcha<br>nalyticsconsulting<br>.com | 6 years of experience working with community partners on research and evaluation | Research<br>Analytics<br>Consulting | Assistant<br>Evaluator |
| Angela<br>Turner | angela.turner@am<br>tcassociates.com | 25+ years of experience consulting for partners from national to local levels, including many projects related to pregnancy prevention and sexual risk avoidance in youth | AMTC | Guiding<br>Evaluator |

## Appendix A. Logic Model

New Jersey Physicians Advisory Group (NJPAG) PREIS Program

#### Program Logic Model (LM)

Target Population: 9th graders in Newark, New Jersey public schools.

NJPAG: Board of Directors. M. Cowan (Executive Director); A. Markarian, MPH, CHES (Program Director); C. Antoine, B. Jerome, I. Antoine, J. Satz (Educators)

Newark Public Schools: Malcolm X Shabazz High School Weequahic High School Bard Early College High School American History High School Newark School of Global Studies Newark Vocational High School University High School West Side High School Arts High School Technology High School

Evaluators: AMTC & Associates: Angela Turner, Immaculate Apchemengich, Melanie Porterfield, Salvador Dominguez, Dr. Cindy Walker, Helena Lucia Swanson

#### 9th Grade Curriculum:

YES You Can...Make Smart Choices!

#### Trained Staff:

By Program Director: Overall program model, curriculum, periodic professional development.

By Evaluation Team: Evaluation/survey protocol.

Approval from Newark, New Jersey Board of Education to deliver curriculum in health classes. Relationship with school staff.

Outcomes Activities Implement Curriculum: YES You Can...Make Smart Choices! Longer Term Outcomes (YYC...MSC!) Lesson 6: Pregnancy Report increased intent to consistently use Goal: Students will understand pregnancy, how to prevent it, and the contraceptives. Report reduced rates of unprotected sex. consequences of pregnancy. Lesson 8: Avoiding Risk Report increased knowledge of HIV/ Goal: Students will understand HIV/AIDs, STDs/ STIs, and unintended Report reduced rates of intent to engage in STDs/STIs. pregnancy, and how to prevent them. sexual activity. proved life skills: Lesson 1: Truth, Dare, or Consequences? · Emotional coping Goal: Students will understand the influences and consequences to sexual Sexual health activity. Report reduced rates of engaging in oral sex. Cognitive Social Lesson 9: What Are We Waiting For? Goal: Students will understand the benefits of refraining from sexual activity. Report increased ability to resist negative Report reduced rates of engaging in sexual Lesson 10: Establishing Healthy Boundaries pressure to have sex. Decreased incidence of pregnancy in target population. Goal: Students will understand personal boundaries and how to resist and refuse sexual activity. Lesson 2: Dare To Be You Goal: Students will understand how others influence their character Decreased incidence of STIs in target population. development and decision-making. Report increased knowledge of healthy relationships. Lesson 3: Intimacy Goal: Students will understand intimacy and when to be intimate in relationships Enhanced character development in target population. Lesson 4: Relationship Health Part 1 Goal: Students will begin to understand what love is and how to have healthy Report increased communication skills. Report increase in future orientation and etting life goals. Lesson 5: Relationship Health Part 2 Goal: Students will continue to understand what love is and know the difference between a healthy and unhealthy relationship. Lesson 11: Effective Communication Goal: Students will understand and obtain skills for effective communication, Report increased financial literacy. including with parents/guardians. Lesson 7: Finances and Future Planning Goal: Students will understand the basics of financial literacy and creating

## Appendix B. Contrast Table

*Note:* The following are constants for all contrasts in the below table:

Design = RCT

Target Population = Youth in 9<sup>th</sup> grade in urban school districts in the Northeast region, without any severe cognitive, mental, or behavioral impairments

Sample Eligibility Criteria: All students enrolled in health classes in participating schools

Treatment Description: Youth receiving YYC...MSC! program

Control Description: Business as usual

Baseline Unit of assignment/observation: Measure [Scale]: The same measurement will be used at baseline and outcome; therefore, only the outcome is detailed in the table

| | Outcome | | |
|---|---|---|---|
| Research Question:<br>Primary/ Secondary | Domain | Unit of assignment/ observation: Measure [Scale] | Timing of measurement |
| RQ 0 – Primary: | | | |
| What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' reports of engaging in sexual intercourse 12-months after the pre-survey compared to those that do not receive the program? | Sexual Activity | Individual participants: Survey – sexual intercourse in the last 3 months. 1-item measure asking participants how many times they engaged in sexual intercourse in the past 3-months recoded to a dummy variable (1 = had sex in the last 3-months, 0 = did not have sex in the last 3-months) | 12-months after pre-survey |
| RQ 1 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in | Sexual Activity | Individual participants: Survey – 8-item<br>Sexual Intimacy Spectrum scale with a 5-<br>point frequency scale | 3-months after pre-survey, 12-months after pre-survey |

| Northeast urban school districts' reports of engaging in oral sex compared to those that do not receive the program? | | Individual participants: Survey – Two 1-<br>item measures asking participants if they<br>ever engaged in oral sex if so, how many<br>times have they done it in the past 3-<br>months | |
|---|---|---|---|
| RQ 2 – Secondary: | | | |
| What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' reports of intent to engage in sexual activity compared to those that do not receive the program? | Intent to Engage in Sexual Activity | 8-item Sexual Initiation scale with a 5-point success sequence response scale Individual participants: Survey – 5-item Intentions to Engage in Sexual Intercourse scale with a 6-point Agree scale | Post-survey, 3 months after pre-<br>survey, 12 months after pre-survey |
| RQ 3 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' reports intent to consistently use contraception compared to those that do not receive the program? | Sexual Risk Avoidance Intent | Individual participants: Survey – Two 1- item measures asking: "If you have sexual intercourse tomorrow, will you make sure a condom is used?" & "If you have sexual intercourse tomorrow, will you make sure birth control is used?" Both questions use the same 5-point response scale: Yes, No, Only if my partner agrees, I don't know/I'm not sure. This question does not apply to me because I do not plan to have sexual intercourse soon Individual participants: Survey – Four 1- item measures asking if youth or their partner have used the following methods in the last month and what they intend to | Post-survey, 3 months after presurvey, 12 months after pre-survey |

| | | | 27 |
|---|---|---|---|
| | | use in the future: condoms, pull-out method, birth control, other contraceptives | |
| RQ 4 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' reports of having unprotected sex compared to those that do not receive the program? | Sexual Risk Avoidance | Individual participants: Survey – If youth mentioned previously having sexual intercourse: In the <b>past 3 months</b> (90 days), how many times did you or your partner use a condom when engaging in sexual intercourse? Response: 0-10+ In the <b>past 3 months</b> (90 days), how many times did you or your partner use the pull-out method when engaging in sexual intercourse? Response: 0-10+ Or I don't know what this is. In the past 3 months, have you or your partner used either of the following methods to prevent pregnancy: 1. Birth control pills 2. Other forms of contraceptive methods, not including a condom (e.g., shot, patch, IUD, etc.). Response options: Yes, No, Unsure | 3 months after pre-survey & 12 months after pre-survey |
| RQ 5 – Secondary: | | | |
| What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' increased financial literacy compared to those that do not receive the program? | Life Skills | Individual participants: Survey – 6-item Financial Literacy scale – 3 items are true/false, and the other 3 are strongly disagree-strongly agree | Post-survey, 3 months after pre-<br>survey, 12 months after pre-survey |

| RQ 6 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' knowledge of HIV/STDs/STIs compared to those that do not receive the program? | Sexual Health Knowledge | Individual participants: Survey – 7-item<br>Knowledge of Sexual Risks scale with<br>True/False/Unsure response scale | Post-survey, 3 months after pre-<br>survey, 12 months after pre-survey |
|---|---|---|---|
| RQ 7 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' reports of their ability to resist negative pressures to have sex compared to those that do not receive the program? | Sexual Risk Avoidance Skills | Individual participants: Survey – 6-item<br>Skills to Resist Pressure (Coercion) to<br>Have Sex scale with a 5-point Confidence<br>response scale | Post-survey, 3 months after pre-<br>survey, 12 months after pre-survey |
| RQ 8 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' reports of future orientation and setting life goals compared to those that do not receive the program? | Life Skills | Individual participants: Survey – 5-item<br>Goal Attainment scale with 6-point Agree<br>response scale | Post-survey, 3 months after presurvey, 12 months after pre-survey |

| | | 1 | 20 |
|---|---|---|---|
| RQ 9 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' reports of healthy life skills compared to those that do not receive the program? | Life Skills | Individual participants: Survey – Combination of all scales except Financial Literacy | Post-survey, 3 months after pre-<br>survey, 12 months after pre-survey |
| RQ 10 – Secondary: | | | |
| What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' knowledge of healthy relationships compared to those that do not receive the program? | Life Skills | Individual participants: Survey – 6-item Awareness of Relationship Safety scale with 6-point strongly disagree-strongly agree response scale Individual participants: Survey – 7-item Dating Choices scale with a 4-point Likelihood response scale | Post-survey, 3 months after pre-<br>survey, 12 months after pre-survey |
| RQ 11 – Secondary: What is the effect of the 2-week YYCMSC! program on 9th grade students in Northeast urban school districts' increased communication skills compared to those that do not receive the program? | Life Skills | Individual participants: Survey – 7-item Communication Scale with a 5-point Confidence scale | Post-survey, 3 months after pre-<br>survey, 12 months after pre-survey |
| RQ 12 – Secondary: | Sexual Activity | Individual participants: Survey – sexual intercourse in the last 3 months. 1-item | 3-months after pre-survey |

| What is the effect of the 2- | measure asking participants how many |
|---|---|
| week YYCMSC! program | times they engaged in sexual intercourse |
| on 9th grade students in | in the past 3-months recoded to a dummy |
| Northeast urban school | variable $(1 = had sex in the last 3-months,$ |
| districts' engaging in sexual | 0 = did not have sex in the last 3-months) |
| intercourse 3-months after | |
| the pre-survey? | |

### Appendix C: Parental Written Notice

# Parent/Guardian Written Notice YES You Can... Make Smart Choices! Evaluation Study

### Introduction

Your child's/student's school has agreed to participate in the evaluation of character development and pregnancy prevention program called *Yes You Can... Make Smart Choices!* The information provided in this written notice is to inform you of what your child/student could participate in.

### What will your child/student be asked to do?

If your child/student participates in the evaluation, they will be asked to:

- Complete an entry survey
- Complete three follow-up surveys 2 weeks after the entry survey, 3 months from the entry survey date, and 12 months from the entry survey date.

### Why is this study being done on this program?

- To:
  - o Determine the impact of the program on participants' attitudes, knowledge, and behaviors.
  - o Collect information that will help:
    - improve the program; and
    - provide the funder, the federal government, with data required on programs they support.

These surveys will address a variety of relationship and sexual health topics, including behaviors, sexual activity, contraception use, and knowledge of STDs/HIV. It will also ask them to provide their demographic information (i.e., gender, race/ethnicity, etc.).

### Will students receive gift cards?

Yes, every student that participates in the survey responses will receive \$20 after completing the second survey, \$30 after the third, and an additional \$40 after completing the 4<sup>th</sup> survey, totaling \$90 over a year's time.

### What are the benefits of the evaluation study?

Students will receive no direct benefits, other than gift cards, for participating in the evaluation study. However, their participation will help the developer of the curriculum, NJ Physicians Advisory Group (NJPAG), determine the impact of the YES You Can...Make Smart Choices! program.

### Are there any risks to students involved in the study?

A potential risk is that some students might find certain questions to be sensitive. Students may skip questions that they do not want to answer. In any study, there is always some risk of a breach of confidentiality. However, the survey has been designed to protect your child's privacy. Students will not put their names on the survey. There will be a confidential ID that links surveys to each other, using their first and last initials and their month and day of birth. However, this information will **only** be accessible to the researchers. Also, no class or student will **ever** be mentioned by name in the final report of the results.

### **Certificate of Confidentiality**

To further protect your child's privacy, the researchers involved in the study have applied for a Certificate of Confidentiality from the National Institutes of Health. Researchers with this certificate agree to keep your child's responses private to the extent permitted by New Jersey law.

### Do students have to participate in this study?

No, this study is voluntary. Parents/guardians may choose to opt their child/student out of the study by completing this form and the student returning it on time. Students may decline to participate or withdraw at any time. They will also be assured that refusing to participate in the evaluation study will not impact their classroom work or grade in any way.

### What if a student does not want to participate in the study?

If a student does not want to participate, then they will not be included in the study, and there will be no penalty.

### Will all students participating in the study have the YES You Can! Program taught?

Not all participating students in this study will be selected to receive the program. Classes will be randomly selected to receive this program, and classes NOT selected for the program will receive alternative lessons and will complete a total of four (4) surveys to receive gift cards, totaling \$90.

How will students' privacy and confidentiality be protected if they decide to participate in this study? Privacy and confidentiality will be protected since students will remain anonymous to NJPAG, parents, and the school district. Survey responses will be stored on the cloud on a password-protected computer and the only people who will have access to individual responses are the researchers, located in another state, who are conducting the evaluation.

If it becomes necessary for an Institutional Review Board to review the study records, information that can be linked to your child will be protected to the extent permitted by law. Your child's research records will not be released without your consent unless required by law or a court order.

### **Future Use of Information**

Even if researchers, not detailed in this consent form, were ever to review the data for research purposes, no data will contain information that could be associated with your child.

### **Clinically Relevant Research Results**

The results of this evaluation study will not be shared with participants.

### Who should I contact with questions about the evaluation study?

Prior, during, or after providing your consent you can contact Dr. Cindy Walker, Consultant for AMTC and Associates (AMTC) at (414) 218-2442. AMTC is the organization responsible for the evaluation of this program. If you have any questions about your child/student's rights, as a participant in this research, or if you feel your child has been placed at risk, you can contact the BRANY IRB Office at (516) 318-6877.

## Parents/guardians, THERE IS <u>NO ACTION NEEDED</u> IF YOU AGREE TO YOUR CHILD/STUDENT PARTICIPATING IN THE EVALUATION STUDY.

| Following New Jersey Bill A5597 (see link below), parents/guardians may opt their child/student out of the evaluation study by checking the box below and telling the student to return this form to their health class before the deadline. |
|---|
| ☐ I would like to opt my child/student out of the evaluation study. |
| Parent's/Guardian's name |
| Child's/Student's name |
| To devile Date |

### Appendix D: Enrollment Form

# New Jersey Physicians Advisory Group (NJPAG) Yes You Can...Make Smart Choices!

### **Enrollment Form**

1. What is your **FIRST NAME**?

2. What is your LAST NAME?

| Note: | Please | write a | as neatly | / as | possible | on | this | form. |
|-------|--------|---------|-----------|------|----------|----|------|-------|

3. How old are you? (MARK ONLY ONE ANSWER)

a. 10b. 11

| | | 12<br>13 |
|---|---|---|
| | | 14 |
| | | 15 |
| | | 16 |
| | | 17 |
| | i. | 18 |
| 4. | Are you Hi | ispanic or Latino? (MARK YES OR NO) |
| | | Yes |
| | b. | No |
| 5. | What is vo | ur race? (MARK ALL THAT APPLY) |
| | - | American Indian or Alaska Native |
| | b. | Asian |
| | | Black or African American |
| | | Native Hawaiian or Other Pacific Islander |
| | | White or Caucasian |
| | f. | Other (specify): |
| 6. | What is yo | our sex? (MARK ONLY ONE ANSWER) |
| | a. | Male |
| | b. | Female |
| sui | rveys. If yo | g for your contact information in the case we need to contact you to participate in follow-up u participate in follow-up surveys you are given a \$30 gift card for the 3-month follow-up, a \$40 he 12-month follow-up survey, and you will be entered into a raffle to win prizes |
| _ | *** | |
| 7. | What is a | reliable phone number you can be reached at via text or call? |
| 8. | What is a | reliable email you can be reached at? |
| | ← CF | IECK THIS BOX IF YOU AGREE FOR US TO TEXT, CALL OR EMAIL YOU IN REGARD |
| | | HE STUDY. |
| | <u> </u> | |

### Appendix E: Survey

### YOUTH ASSENT FORM

You are being asked to participate in the evaluation of the New Jersey Physician Advisory Group *Yes You Can...Make Smart Choices!* program by completing the following questionnaire. The program is designed to teach youth about pregnancy prevention and further their character development. This evaluation will help to improve and ensure the program is interesting and helpful. Upon receiving parental consent, youth will be asked to participate in four (4) data collection periods.

Your participation in this survey is voluntary, meaning you do not have to participate if you do not want to.

Some of the questions that you will be asked are personal. We hope that you will answer all of the questions, but you may skip any questions you do not wish to answer.

The answers you give will be kept private to the extent permitted by law. This means that none of your responses will be shared with any of your teachers, or anyone at your school, or any of your family and friends. The only person who will have access to your responses are external consultants. In addition, no one will report any individual responses to this survey - we will only report on the combined responses across all of the students that take part in the *Yes You Can...Make Smart Choices!* program.

Thank you!

Do you agree to participate in the evaluation?

- a. Yes (Continue to Performance Measures)
- *b.* No (*Skip to END OF SURVEY*)

### THE PAPERWORK REDUCTION ACT OF 1995

Public reporting burden for this collection of information is estimated to average 16 minutes per response, including the time for reviewing questions, gathering and maintaining the data needed, and reviewing the collection of information. An agency may not conduct or sponsor, and a person is not required to respond to, a collection of information unless it displays a currently valid OMB control number. The information collected will help policy makers and other stakeholders understand the experiences of youth today and identify ways to reduce risky behaviors. The information will also inform programs on how best to serve their participants. The collection of information is voluntary, and responses will be kept private to the extent allowed by law. THE OMB number for this information collection is 0970-0497 and the expiration date is 06/30/2023.

| PLEASE READ EACH QUESTION CAREFULLY: There are different ways to answer the questions in |
|---|
| this survey. It is important that you follow the instructions when answering each kind of question. Here |
| are some examples |

| 1 | $\mathbf{E}\mathbf{X}$ | AN | ЛPI | $\mathbf{E}$ | 1 • | $\mathbf{M}$ | ARK | ONLY | ONE | <b>ANSWER</b> |
|---|---|---|---|---|---|---|---|---|---|---|
| | 17/ | | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | 1 1 | | | 71717 | 171111 | | |

What is the color of your eyes?

If the color of your eyes is brown, you would mark (X) the first box as shown.

### MARK ONLY ONE ANSWER

| $\boxtimes$ | Brown |
|-------------|---------------|
| | Blue |
| | Green |
| | Another color |

### 2. EXAMPLE 2: MARK ALL THAT APPLY

Do you plan to do any of the following next week?

### MARK ALL THAT APPLY

☑ Watch a movie

If you plan to watch a movie <u>and</u> go to a baseball game next week, you would mark both boxes.

oxdiv Go to a baseball game

☐ Study at a friend's house

| 1. | How old are you? (MARK ONLY ONE ANSWER) a. 10 b. 11 c. 12 d. 13 e. 14 f. 15 g. 16 h. 17 i. 18 j. 19 k. 20 l. 21 |
|---|---|
| 2. | What grade are you in? (If you are currently on vacation or in summer school, indicate the grade you will be in when you go back to school.) (MARK ONLY ONE ANSWER) a. 5 <sup>th</sup> b. 6 <sup>th</sup> c. 7 <sup>th</sup> d. 8 <sup>th</sup> e. 9 <sup>th</sup> f. My school does not assign grade levels g. I dropped out of school, and I am working on getting a high school diploma or GED h. I am working toward a GED i. I have a high school diploma or GED, but I am <u>not</u> currently enrolled in college or technical school j. I have a high school diploma or GED and I <u>am</u> currently enrolled in college or technical school |
| 3. | When you are home or with your family, what language or languages do you usually speak? (MARK ALL THAT APPLY) a. English b. Spanish c. Other (please specify): |
| 4. | Are you Hispanic or Latino? (MARK YES OR NO) a. Yes b. No |
| 5. | What is your race? (MARK ALL THAT APPLY) a. American Indian or Alaska Native b. Asian c. Black or African American d. Native Hawaiian or Other Pacific Islander e. White or Caucasian f. Other (specify): |
| 6. | What is your sex? (MARK ONLY ONE ANSWER) a. Male b. Female |

7. Are you currently...? (MARK ALL THAT APPLY)

- a. Living with family [parent(s), guardian, grandparents, or other relatives]
- b. In foster care, living with a family
- c. In foster care, living in a group home
- d. Couch surfing or moving from home to home
- e. Living outside in a tent city or homeless camp, in a car, in an abandoned vehicle or in an abandoned building
- f. Staying in an emergency shelter or transitional living program
- g. Staying in a hotel or motel
- h. In juvenile detention center, juvenile group home, and/or under the supervision of a probation office
- i. None of the above

For questions 8-12, please think about how the program you just completed has affected you.

8. Even if your program didn't cover this topic, would you say that being in the program made you more likely, about the same or less likely to... (*Note: If the program has not affected your likelihood to do the following, choose "About the same"*.)

### MARK ONLY ONE ANSWER PER ROW.

| | Much<br>more<br>likely | Somewhat<br>more<br>likely | About the same | Somewhat less likely | Much less likely |
|---|---|---|---|---|---|
| aresist or say no to peer pressure? | | | | | |
| bmanage your emotions in healthy ways (for example, ways that are not hurtful to you or others)? | | | | | |
| cmake decisions to not use drugs and alcohol? | | | | | |
| dthink about the consequences before making a decision? | | | | | |

9. Even if your program didn't cover this topic, would you say that being in the program made you more likely, about the same or less likely to... (*Note: If the program has not affected your likelihood to do the following, choose "About the same".*)

### MARK ONLY ONE ANSWER PER ROW.

| | Much<br>more | Somewhat more | About the | Somewhat less likely | Much<br>less |
|---|---|---|---|---|---|
| | likely | likely | same | | likely |
| amake plans to reach your goals? | | | | | |
| bcare about doing well in school? | | | | | |
| cgraduate high school or get your GED? | | | | | |
| dget more education or training after<br>high school or completing your GED? | | | | | |
| eget a steady full-time job after school? | | | | | |

10. Even if your program didn't cover this topic, would you say that being in the program made you more likely, about the same or less likely to... (*Note: If the program has not affected your likelihood to do the following, choose "About the same"*.)

### MARK ONLY ONE ANSWER PER ROW.

| | Much more likely | Somewhat more likely | About the | Somewhat less likely | Much less likely |
|---|---|---|---|---|---|
| | | | same | | |
| asave money to get things you want? | | | | | |
| bfeel confident about how to open a bank account? | | | | | |
| cfeel confident about how to prepare a budget? | | | | | |
| dfeel confident about how to track your expenses? | | | | | |
| eunderstand the costs associated with raising a child? | | | | | |

11. Even if your program didn't cover this topic, would you say that being in the program made you more likely, about the same or less likely to... (*Note: If the program has not affected your likelihood to do the following, choose "About the same".*)

### MARK ONLY ONE ANSWER PER ROW.

| | Much<br>more<br>likely | Somewhat more likely | About the same | Somewhat less likely | Much<br>less<br>likely |
|---|---|---|---|---|---|
| atalk with your parent, guardian, or caregiver about things going on in your life? | | | | | |
| btalk with your parent, guardian, or caregiver about sex? | | | | | |

12. Even if your program didn't cover this topic, would you say that being in the program made you more likely, about the same or less likely to... (*Note: If the program has not affected your likelihood to do the following, choose "About the same"*.)

### MARK ONLY ONE ANSWER PER ROW.

| | Much | Somewhat | About the | Somewhat | Much less |
|---|---|---|---|---|---|
| | more | more | same | less likely | likely |
| | likely | likely | | | |
| abetter understand what makes a relationship healthy? | | | | | |

| bresist or say no to someone if they pressure you to participate in sexual acts, such as kissing, touching private parts, or sex? |
|---|
| ctalk to a trusted person/adult (for example, a family member, teacher, counselor, coach, etc.) if someone makes you uncomfortable, hurts you, or pressures you to do things you don't want to do? |

The next questions ask about sexual intercourse.

- 13. As a result of being in the program, are you planning to abstain from sexual intercourse (choose to not have sexual intercourse) for at least the next 3 months?
  - a. Yes (Skip to Question 14)
  - b. No (Skip to Question 15)
  - c. Not sure (Skip to Question 15)
- 14. How important are each of these reasons for your decision to not have sexual intercourse for at least the next 3 months? MARK ONLY ONE ANSWER PER ROW.

| | Not at all | Not too | Somewhat | Very |
|---|---|---|---|---|
| | important | important | important | important |
| ahow it might affect your plans for the future? | | | | |
| bthe possible emotional and social consequences | | | | |
| (for example, feeling sadness or regret, | | | | |
| disappointing your parent(s) or guardian(s), and/or | | | | |
| negative reactions from your peers)? | | | | |
| cthe risk of getting a sexually transmitted infection | | | | |
| (STI)? | | | | |
| dthe risk of getting pregnant or getting someone | | | | |
| pregnant? | | | | |



IF YOU ANSWERED "YES" TO QUESTION 13, GO TO QUESTION 14

IF YOU ANSWERED "NO" OR "NOT SURE" TO QUESTION 13: SKIP QUESTION 14 AND GO TO QUESTION 15 ON THE NEXT PAGE
15. The next few questions refer to sexual intercourse and your risk of pregnancy and sexually transmitted infections (STIs). Remember, all your responses will be kept private.

Has being in the program made you more likely, about the same, or less likely to... (*Note: If the program has not affected your likelihood to do the following, choose "About the same"*.)

- a. ...have sexual intercourse in the next 3 months? MARK ONLY ONE ANSWER.
  - a. Much more likely
  - b. Somewhat more likely
  - c. About the same
  - d. Somewhat less likely
  - e. Much less likely
- b. ...use (or ask your partner to use) a condom if you were to have sexual intercourse in the next 3 months? MARK ONLY ONE ANSWER.
  - a. This question does not apply to be because I choose to not have sexual intercourse in the next 3 months
  - b. Much more likely
  - c. Somewhat more likely
  - d. About the same
  - e. Somewhat less likely
  - f. Much less likely
- c. ...use (or ask your partner to use) birth control OTHER than condoms if you were to have sexual intercourse in the next 3 months? By birth control, we mean methods that can prevent pregnancy, like using birth control pills, the shot, the patch, the ring, IUD, or implant.
  - a. This question does not apply to be because I choose to not have sexual intercourse in the next 3 months
  - b. Much more likely
  - c. Somewhat more likely
  - d. About the same
  - e. Somewhat less likely
  - f. Much less likely

16. The next questions ask you about your experiences in the program that you just completed. Think about all the sessions or classes of the program that you attended.

Even if you didn't attend all sessions or classes in this program, how often in this program...

## MARK ONLY ONE ANSWER PER ROW.

| | All of the time | Most of the time | Some of the time | None of the time |
|---|---|---|---|---|
| adid you feel interested in program sessions and | | | | |
| classes? | | | | |
| bdid you feel the material presented was clear? | | | | |
| cdid the discussions or activities help you learn | | | | |
| program lessons? | | | | |
| ddid you have a chance to ask questions about topics | | | | |
| or issues that came up in the program? | | | | |
| edid you feel respected as a person? | | | | |

17. Thinking about the program, how satisfied are you with...

#### MARK ONLY ONE ANSWER PER ROW.

| | Very | Somewhat | A little | Not at |
|---|---|---|---|---|
| | satisfied | satisfied | satisfied | all |
| | | | | satisfied |
| athe amount of information you received about | | | | |
| abstaining from sex (choosing to not have sex)? | | | | |
| bthe amount of information you received about | | | | |
| condoms and birth control? | | | | |

#### **DEMOGRAPHICS**

# The following questions allow us to link the pre-, post-, and follow-up surveys to provide more confidentiality for you.

What is the first letter in your **first** name? (Example: **J** ohn)

(Drop down with A-Z)

What is the first letter in your **last** name? (Example: S mith)

(Drop down with A-Z)

What is the **month** of your birthday?

(Drop down with Jan-Dec)

What **day** of the month is your birthday?

(Drop down with 1-31)

#### The following questions will be used to help us describe whom the program is serving.

What gender do you identify with?

- a. Boy
- b. Girl
- c. Non-binary/ Gender-fluid

Do you identify as transgender?

- a. Yes
- b No
- c. I am not sure
- d. I do not know what this question is asking

Which of the following best describes you?

- a. Heterosexual (straight)
- b. Gay or lesbian
- c. Bisexual
- d. I am not sure about my sexual identity (questioning)
- e. I do not know what this question is asking
- f. None of the above

Are you in a romantic relationship right now (e.g., going out or hanging out with someone)?

- a. Yes
- b. No
- c. Unsure/It's complicated

Were you in a romantic relationship at any point in the last 3-months?

- a. Yes
- b. No
- c. Unsure/It's complicated

In the past 12 months, have you learned about any of the following topics in a school or other formal learning setting (e.g., Boys and Girls Club, church)?

| | Yes | No |
|-------------------------------------------------------------|-----|----|
| a. Relationships, dating, or marriage | | |
| b. Waiting until you are ready to engage in sexual activity | | |
| c. Methods of birth control, such as condoms, pills, etc. | | |
| d. Sexually transmitted diseases also known as STDs or STIs | | |
| e. Communication | | |
| f. Financial literacy | | |

### PROGRAM SATISFACTION QUESTIONS

The next two questions ask you to reflect on your experiences while taking the program.

How likely are you to recommend this program to a friend?

- a. Not at all likely
- b. Somewhat likely
- c. Likely
- d. Very likely

What is the best thing you learned about yourself in the program? [OPEN-ENDED]

#### **COMMUNICATION SKILLS**

How CONFIDENT are you that you could do each of the following things:

| | Not at all confident | A little confident | Somewhat confident | Confident | Completely confident |
|---|---|---|---|---|---|
| Show that you care about someone else's feelings. | | | | | |
| Calmly explain how you feel. | | | | | |
| Suggest a compromise to end an argument. | | | | | |

| Agree to try a solution someo suggested to end an argument | | | | |
|---|---|---|---|---|
| Clearly communicate your the someone else. | oughts to | | | |
| Listen carefully to what some telling you. | one else is | | | |
| Show that you care about som opinion. | neone else's | | | |
| DATING CHOICES | | | | |
| Thinking of yourself right now | how likely are you to | date someone who | ` | |
| Thinking of yourself right now | , how likely are you to Not at all likely | date someone who<br>Somewhat<br>likely | Likely | Very likely |
| Thinking of yourself right now is <b>much</b> older than you. | | Somewhat | | Very likely |
| | | Somewhat | | Very likely |
| is <b>much</b> older than you keeps you a secret from | Not at all likely | Somewhat | | Very likely |
| is <b>much</b> older than you. keeps you a secret from others. calls you names when they | Not at all likely | Somewhat | | Very likely |
| is <b>much</b> older than you. keeps you a secret from others. calls you names when they are upset. | Not at all likely | Somewhat | | Very likely |
| is <b>much</b> older than you. keeps you a secret from others. calls you names when they are upset. respects your boundaries. | Not at all likely | Somewhat | | Very likely |

## AWARENESS OF RELATIONSHIP SAFETY

How much do you agree with each of the following statements.

| | Strongly<br>Disagree | Disagree | Somewhat<br>Disagree | Somewhat<br>Agree | Agree | Strongly<br>Agree |
|---|---|---|---|---|---|---|
| If my partner ever hit me, we would have to break up. | | | | | | |
| If I were afraid of my partner, I would know where to go for help. | | | | | | |
| It is acceptable for me to hit my partner if I am angry. | | | | | | |
| I would end a relationship with someone if they tried to force me to do things I didn't want to do. | | | | | | |
| If my partner <b>always</b> tried to tell me what to do, we would have to break up. | | | | | | |
| I would stay with my partner if they called me names and put me down, as long as they said they love me. | | | | | | |

## KNOWLEDGE OF SEXUAL RISKS

Pick either True, False, or Unsure for the following questions:

| | True | False | Unsure |
|---|---|---|---|
| A girl can get pregnant the first time she has unprotected vaginal sexual intercourse. | | | |
| Using a condom will always prevent a sexually transmitted disease/infection (STD/STI) | | | |
| A person with NO symptoms can still spread an STD/STI through sexual activity. | | | |
| The only sure way to prevent pregnancy is to avoid sexual activity. | | | |
| A person can get an STD/STI from oral sex. | | | |
| The only way to prevent an STD/STI is to avoid sexual activity. | | | |
| If someone has unprotected sexual intercourse, even once, they can get an STD/STI like HIV. | | | |

# SKILLS TO RESIST PRESSURE (COERCION) TO HAVE SEX

How CONFIDENT are you that you could do each of the following?

| | Not at all confident | A little confident | Somewhat confident | Confident | Completely confident |
|---|---|---|---|---|---|
| Avoid situations that could lead to unwanted sexual activity (like being alone with someone in a bedroom). | | | | | |
| Avoid people who make you feel pressured to have sexual intercourse. | | | | | |
| Firmly say "no" to sexual activity, even if someone is pressuring you. | | | | | |
| Firmly say "no" to your partner if you do not want to have sexual intercourse. | | | | | |
| End a relationship with someone pressuring you to have sexual intercourse when you do not want to. | | | | | |
| Wait until you are ready to have sexual intercourse. | | | | | |

## SEXUAL INTIMACY SPECTRUM

In the following items, we are talking about voluntary intimate/ sexual activity.

In the past month, how often have you engaged in these intimate activities with a romantic partner?

| | Never | A few times in the last month | Once a week | A few times a week | Daily |
|---|---|---|---|---|---|
| Kissing | | | | | |
| Spending time alone together in a private space (e.g., bedroom) | | | | | |
| Laying down together | | | | | |
| Sexting (e.g., sending, receiving, or forwarding sexually explicit messages, photographs, or videos digitally via mobile phones or through social media) | | | | | |
| Touching under clothing Oral sex | | | | | |
| Sexual intercourse | | | | | |
| Other sexual activity (please specify): | | | | | |

# SEXUAL INITIATION

When do you think you may engage in each of the following activities:

| | Within the next<br>12 months | Before<br>graduating<br>high school | After graduating high school | After starting a career | After an adult committed relationship, like marriage |
|---|---|---|---|---|---|
| Kissing | | | | | |
| Spending time alone together in a private space (e.g., bedroom) | | | | | |
| Laying down together | | | | | |
| Sexting (e.g., sending, receiving, or forwarding sexually explicit messages, photographs, or videos digitally via mobile phones or through social media) | | | | | |
| Touching under clothing | | | | | |
| Oral sex | | | | | |
| Sexual intercourse | | | | | |
| Other sexual activity (please specify): | | | | | |

#### INTENTIONS TO ENGAGE IN SEXUAL INTERCOURSE

Indicate your level of agreement with each of the following statements:

| | Strongly disagree | Disagree | Somewhat Disagree | Somewhat<br>Agree | Agree | Strongly<br>Agree |
|---|---|---|---|---|---|---|
| Engaging in sexual intercourse at this time could prevent me from reaching my goals. | | | | | | |
| Engaging in sexual intercourse right now is probably not a good idea. | | | | | | |
| I think it's a good idea to finish high school before engaging in sexual intercourse. | | | | | | |
| I am strongly committed to wait until marriage to have sexual intercourse. | | | | | | |
| I do not plan to have sexual intercourse any time soon. | | | | | | |

#### INTENT TO CONSISTENTLY USE CONDOMS

If you have sexual intercourse tomorrow, will you make sure a condom is used?

- a. Yes
- b. No
- c. Only if my partner agrees
- d. I don't know / I'm not sure
- e. This question does not apply to me because I do not plan to have sexual intercourse soon.

If you have sexual intercourse tomorrow, will you make sure birth control is used?

- a. Yes
- b. No
- c. Only if my partner agrees
- d. I don't know / I'm not sure
- e. This question does not apply to me because I do not plan to have sexual intercourse soon.

#### SEXUAL ACTIVITY

In the following items, we are talking about voluntary intimate/ sexual activity.

[Qualifying question]: Have you ever had oral sex? Response: Y/N

[Branch questions if Y to previous question, Qualifying question]:

In the past 3 months (90 days), how many times have you had oral sex? Response:0-10+

[Qualifying question]: Have you ever had sexual intercourse? Response: Y/N

[Branch question if Y to previous question, Qualifying question]:

In the **past 3 months** (90 days), how many times have you had sexual intercourse? Response: 0-10+

#### CONDOM & CONTRACEPTIVE USAGE

[Branch section if more than 0 to the following question: In the **past 3 months** (90 days), how many times have you had sexual intercourse?]

There are different types of contraceptives that may be used including condoms, birth control pills, the pull-out method, and other contraceptives (e.g., shot, patch, IUD, etc.).

In the **past 3 months** (90 days), how many times did you or your partner use a condom when engaging in sexual intercourse? Response: 0-10+

In the **past 3 months** (90 days), how many times did you or your partner use the pull-out method when engaging in sexual intercourse?

Response:

0 - 10 +

I don't know what this is.

In the **past 3 months**, have you or your partner used either of the following methods to prevent pregnancy:

| _ | Yes | No | Unsure |
|---|---|---|---|
| Birth control pills | | | |
| Other forms of contraceptive methods, not including a condom (e.g., shot, patch, IUD, etc.) | | | |

## GOAL ATTAINMENT

How much you agree with each of the following statements:

| | Strongly<br>Disagree | Disagree | Somewhat<br>Disagree | Somewhat<br>Agree | Agree | Strongly<br>Agree |
|---|---|---|---|---|---|---|
| I know how to set goals. | | | | | | |
| I know what I want for my future. | | | | | | |
| I know what steps to take to achieve my goals. | | | | | | |
| If I or my partner were to become pregnant now, it <b>could</b> prevent me from reaching my long-term goals. | | | | | | |
| I know I can reach my long-term goals, even if challenges occur. | | | | | | |
| NANCIAL LITERACY | | г.1 | T.I. | | | |

## FIN

Please respond to the following questions with either True, False, or Unsure.

| | True | False | Unsure |
|---|---|---|---|
| When you use a debit card, you are <b>borrowing</b> money from the bank that you must pay back. | | | |
| Missing only one credit card payment will impact your credit score. | | | |
| I understand the difference between credit cards and debit cards. | | | |

Please respond to the following questions:

| Strongly<br>Disagree | Disagree | Somewhat Disagree | Somewhat Agree | Agree | Strongly<br>Agree |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

I know how to create a budget for earning, spending, and saving my money.

I am too young to start thinking about budgeting my money.

I know how to set financial goals.

## **END OF SURVEY**

Thank you!